CLINICAL TRIAL: NCT05274828
Title: Feasibility Study on the Use of an Intensive Deep Transcranial Magnetic Stimulation Protocol in the Treatment of Cocaine and Other Stimulants Use Disorder
Brief Title: Deep Transcranial Magnetic Stimulation for Stimulants Use Disorder
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Centre hospitalier de l'Université de Montréal (CHUM) (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 21.358
Record Dates: First submitted 2022-02-16; First posted 2022-03-11 (Actual); Last update posted 2024-04-17 (Actual); Status verified 2024-04

CONDITIONS: Stimulants Use Disorder

STUDY DESIGN:
Intervention Model Description: Single Group Assignment
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- H7-Coil Deep TMS Treatment (Experimental): H7-Coil Deep TMS Treatment
  Interventions: Device: H7-Coil Deep TMS for CUD

INTERVENTIONS:
Device: H7-Coil Deep TMS for CUD — The Study group will receive dTMS treatment three times a day for ten days.
  Other Names: H7-Coil Deep TMS Treatment

SUMMARY:
The purpose of the study is to explore the Feasibility, Tolerability and Safety of the H7-Coil deep Transcranial Magnetic Stimulation for Subjects with Stimulants Use Disorder (SUD).

DETAILED DESCRIPTION:
Stimulants Use Disorder (SUD) is a major public health issue, with potentially severe psychosocial and medical consequences. Even though psychosocial therapies exist, an important proportion of patients do not respond to these approaches, and no approved biological approaches are currently available. deep TMS (dTMS) has been shown effective for Major Depressive Disorder, Obsessive Compulsive Disorder and Nicotine Use Disorder and could also prove available for SUD. Several pilot studies have shown preliminary effectiveness in SUD, but are limited by the length of their protocol, which could result in limited real-world effectiveness secondary to high dropout rates. Given that aTMS protocols have been applied successfully in MDD, we propose to implement this approach for SUD, in order to reduce treatment length and therefore increase retention rates. We will also gather preliminary data on various biomarkers that could help predict response and better understand biological mechanisms behind SUD.

ELIGIBILITY:
Inclusion Criteria:

* Being diagnosed with SUD (moderate or severe) based on DSM-5 criteria
* Current stimulants use with last use in the two weeks prior to admission to the study as confirmed by the Timeline Followback Questionnaire
* Wanting to stop the intake of stimulants
* Being able and willing to adhere to the treatment schedule
* Filling the criteria of the TMS adult safety screening (TASS) questionnaire
* Being voluntary and competent to consent to treatment
* Ability to speak and read French or English

Exclusion Criteria:

* Severe psychiatric condition (history of schizophrenia, schizoaffective disorder or bipolar disorder); current acute psychosis, mania or active suicidality (unipolar major depression, anxiety disorders and personality disorders will be allowed as long as they are not primary and causing greater impairment than SUD)
* Severe and/or unstable medical illness, including but not limited to any neurologic, cardiac, renal or hepatic condition
* Implanted medical device (including but not limited to intracranial implants, cardiac pacemaker, medication pump, etc.) or intracranial implant (e.g., aneurysm clips, shunts, stimulators, cochlear implants, or electrodes) or any other metal object within or near the head, excluding the mouth, that cannot be safely removed
* Clinically significant laboratory abnormality, in the opinion of the principal investigator
* Pregnancy or breastfeeding
* Another current severe substance use disorder (except nicotine)
* Anti-craving medication and other psychotropic medications are allowed, but need to have been stable for four (4) weeks before screening
* Currently taking more than lorazepam 2 mg daily (or equivalent) or any dose of an anticonvulsant due to the potential to limit TMS efficacy.
* Non-correctable clinically significant sensory impairment (i.e., cannot hear well enough to cooperate with the interview)

Ages: 21 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Actual)
Dates: Start 2022-11-02 (Actual); Primary Completion 2023-12-31 (Actual); Study Completion 2024-04-01 (Actual)

PRIMARY OUTCOMES:
Feasibility-related endpoints - adherence to dTMS | after 10 days of treatment sessions
  Number of completer treatment sessions
Feasibility-related endpoints - retention rates | after 10 days of treatment sessions
  Number of patients who did not completed the total (40) sessions
Adverse Events reported | up to three months after end of the treatment
  Adverse events reported

SECONDARY OUTCOMES:
Percentage of Positive Urine Drug Screen to Stimulants | up to three months after end of the treatment
  Presence of Stimulants in the Drug Screen Panel
Percentage change on Stimulants Craving Questionnaire | T0 (week 0), T1 (end of treatment, week 2), T2 (week 4), T3 (week 6), T4 (week 14)
  Percentage change on Stimulants Craving Questionnaire
Percentage change on Stimulants Selective Severity Assessment | T0 (week 0), T1 (end of treatment, week 2), T2 (week 4), T3 (week 6), T4 (week 14)
  Percentage change on Stimulants Selective Severity Assessment (Minimum score 0 and Maximum score 126, higher score means worse outcome in terms of substance withdrawal symptoms)
Percentage change on Patient Health Questionnaire (PHQ-9) | T0 (week 0), T2 (week 4), T3 (week 6), T4 (week 14)
  Percentage change on Patient Health Questionnaire (PHQ-9)
Percentage change on General Anxiety Disorder (GAD-7) | T0 (week 0), T2 (week 4), T3 (week 6), T4 (week 14)
  Percentage change on General Anxiety Disorder (GAD-7)

CONTACTS AND LOCATIONS:
Overall Officials: Jean-Philippe Miron, MD, Principal Investigator — Centre hospitalier de l'Université de Montréal (CHUM)
Locations (1):
- Centre Hospitalier de l'Université de Montréal, Montreal, Quebec, Canada

IPD SHARING:
Plan to Share IPD: No